CLINICAL TRIAL: NCT02179814
Title: Neuronal Correlates of Catecholamine Depletion in Patients With Bulimia Nervosa Off Medication and Healthy Controls
Brief Title: Neural Response to Catecholamine Depletion in Subjects Suffering From Bulimia Nervosa in Their Past and Healthy Controls
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Conduct of the first analyses
Sponsor: University of Bern (Other)
Collaborators: Insel Gruppe AG, University Hospital Bern (Other); University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: 132/10; 2011DR1011 (Other: Swissmedic); 32003B_138264 / 1 (Other Grant/Funding Number: SNF)
Record Dates: First submitted 2014-06-25; First posted 2014-07-02 (Estimated); Last update posted 2019-01-24 (Actual); Status verified 2019-01

CONDITIONS: Bulimia Nervosa; Eating Disorders; Dopamine; Reward; Catechol-O-methyltransferase
Keywords: bulimia nervosa; dopamine; reward; catechol-O-methyltransferase; gene; catecholamines; alpha-methyl-para-tyrosine; magnetic resonance imaging
MeSH Terms: conditions — Bulimia Nervosa; Feeding and Eating Disorders | interventions — alpha-Methyltyrosine; Diphenhydramine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- AMPT (Experimental): Experimental:
  alpha-methyl-paratyrosine (AMPT, trade name: Demser), body-weight adjusted dosage (40 mg/kg body weight, maximum 4000mg) at 4 time points over 24 hours
  Interventions: Drug: AMPT/ Demser
- Diphenhydramine & placebo (Sham Comparator): Diphenhydramine (25mg, trade name in Switzerland: Benocten) at the first medication intake time point, placebo at the second to fourth intake time point (medication intake over 24 hours)
  Interventions: Drug: Diphenhydramine; Drug: Placebo

INTERVENTIONS:
Drug: AMPT/ Demser — alpha-methyl-paratyrosine (AMPT, trade name: Demser) body-weight adjusted dosage (40 mg/kg body weight, maximum 4000mg) at 4 medication intake time points over 24 hours
  Arms: AMPT
Drug: Diphenhydramine — Diphenhydramine (25mg) at the first medication intake time point
  Other Names: Benocten (trade name in Switzerland)
  Arms: Diphenhydramine & placebo
Drug: Placebo — Placebo at the second, third and fourth medication intake time point
  Arms: Diphenhydramine & placebo

SUMMARY:
Bulimia nervosa is a severe psychiatric disorder characterized by recurrent binge eating episodes followed by inappropriate compensatory behavior to prevent weight gain such as self-induced vomiting. With this project, the investigators want to investigate the role of the neurotransmitter dopamine in bulimia nervosa. Dopamine is reported to have an important influence on the neural reward system and is involved in the processing of gains and losses. The reward system is functionally connected to the individual perception of rewards in the environment. A previous study revealed that under catecholamine depletion including dopamine depletion women suffering from bulimia nervosa in their past reported mild bulimic symptoms and their reward processing became dysfunctional: their ability to use rewarding stimuli for task solving was diminished.

The aim of this study is to investigate the role of reduced dopamine availability in the development or maintaining of bulimia nervosa and in the dysfunctional processing of rewarding stimuli and negative visual information. Therefore, the investigators hypothesize that catecholamine depletion achieved by oral administration of alpha-methyl-paratyrosine (AMPT) will induce mild bulimic symptoms in females suffering from bulimia nervosa in their past. In addition, they will reveal dysfunctions in reward and emotional processing under catecholamine depletion. Using functional magnetic resonance imaging, the investigators propose that a reduced activation of the nucleus accumbens, a neural structure of the reward system, will be the neural correlate of this dysfunctional reward processing. Furthermore, the amygdala, a neural structure that is involved in emotional processing, will show a higher activation under catecholamine depletion. Genetic factors additionally have an influence on the dopaminergic system. Therefore, the investigators hypothesize that genetic factors, for example the COMT val-158-met polymorphism may have an effect on the behavioral and neural response to catecholamine depletion. In sum, this investigation may help to understand which changes in reward and emotional processing may lead to a reoccurrence of bulimic symptoms.

In future, the findings of this study may help to develop individual pharmacological and psychotherapeutical interventions to enhance the outcome of treatment.

DETAILED DESCRIPTION:
Background

The Monoamine Deficiency Hypothesis is one of the most solid theories of the neurobiology of mood, anxiety disorder, and addiction. There is increasing evidence that monoamine deficiency also plays an important role in bulimia nervosa. Many indications revealed a disturbance of the catecholamine system in bulimia nervosa. In symptomatic bulimic patients, the concentration of norepinephrine and dopamine in cerebrospinal fluid and peripheral blood was lower than in healthy controls. The neurotransmitter dopamine is thought to be importantly involved in the processing of rewarding stimuli.

One instructive paradigm for investigating the relationship between catecholaminergic function and psychiatric disorders has involved the behavioral response to catecholamine depletion achieved by oral administration of alpha-methyl-paratyrosine (AMPT). This medication is a tyrosine hydroxylase inhibitor and, therefore, it reduces availability of catecholamines in the brain by depleting central norepinephrine and dopamine stores. A relatively large interindividual variation in the response to catecholamine depletion has been consistently observed. Genetic factors may conceivably contribute to this variation. The COMT val-158-met polymorphism was found to play a critical role for the activity of the enzyme catechol-O-methyltransferase (COMT) that metabolizes catecholamines after they have been released into the synaptic cleft. The enzyme activity in individuals homozygous for the val-158 allele is about 40% higher than in homozygotes of the met-158 allele. A high activity of this enzyme is thought to be associated with a higher reduction of catecholamines, particularly of dopamine in the prefrontal cortex.

In a previous study Gregor Hasler and colleagues were the first to use catecholamine depletion to evaluate the roles played by norepinephrine and dopamine in the pathophysiology of bulimia nervosa. The results of this study revealed that under catecholamine depletion remitted bulimic participants showed dysfunctions in motivated behavior in a reward task. In addition this study provided preliminary evidence that COMT val-158-met polymorphism explains some of the variance in the behavioral response to catecholamine depletion. However, in eating disorders, the pathway leading from genetic polymorphism to neural activity to neuropsychological abnormalities to risk of eating disorders remains to be determined.

With this new study the investigators want to investigate the neural substrate of the induced bulimia-associated neuropsychological abnormalities with functional magnetic resonance imaging (fMRI). An additional goal is to examine the effect of the COMT val-158-met polymorphism on neural activity.

In the following the investigators will present their central hypotheses:

1. Remitted bulimic participants will reveal impairments in motivated behavior and abnormal neural activation in a reward task following catecholamine depletion.
2. Remitted bulimic participants will show increased amygdala activation during encoding of negative pictures under catecholamine depletion.
3. Participants with homozygous val-158 alleles of the COMT val-158-met polymorphism will show an increased activation in the ventral striatum during a reward task.
4. Participants with at least one met-158 allele of the COMT val-158-met polymorphism will show higher amygdala activation during the encoding of negative emotional visual information.

Objective

This study will further elucidate the etiology and pathophysiology of bulimia nervosa at various levels, ranging from the role of a specific genetic factor to the activity of specific neural networks to neuropsychological abnormalities and clinical symptoms. It may provide important insights into a specific pathogenetic pathway of bulimia nervosa related to the catecholaminergic in particular to the dopaminergic neurotransmitter system. Since a range of drugs targeting this neurotransmitter system are available, this study may directly inform the development of novel therapeutic strategies tailored to individual patients.

Methods

Remitted bulimic and healthy control participants will be enrolled into a double-blind, placebo-controlled cross-over catecholamine/sham depletion study.

The initial assessment comprises physical examinations, a structured psychiatric interview, clinical ratings and neuropsychological testing.

Catecholamine depletion will be induced by administration of AMPT over 24 hours. Sham depletion includes diphenhydramine at the first medication intake time point because AMPT mostly induce mild sedation.

Based on previous reports, the investigators expect maximal depletion 30 hours after the first dose AMPT. Blood samples will be taken at that time to measure serum prolactin levels as a proxy of catecholamine synthesis. Behavioral experiments (tasks assessing reward and emotional processing) will be conducted in a MR-scanner. The participants will complete various self-report ratings before the first, during and after medication intake.

ELIGIBILITY:
Inclusion Criteria:

* female
* age: 18-60
* caucasian ethnicity
* right handedness
* normal or corrected to normal vision and hearing performance
* remitted bulimic participants: have met the DSM IV criteria for bulimia nervosa in the past
* remitted bulimic participants: have been asymptomatic for at least1 month
* signed written informed consent

Exclusion Criteria

* healthy volunteers: any lifetime psychiatric diagnosis
* healthy volunteers: any lifetime psychiatric diagnosis in first-degree relatives
* no or impaired understanding of the tasks or the risks of the study
* medical or neurological illnesses likely to affect physiology or anatomy
* suicidal ideation or suicide attempts within the last 8 weeks
* current use of psychotropic drugs
* history of drug including alcohol and nicotine (not more than 10 cigarettes per day) abuse within 1 year or a lifetime history of alcohol or drug dependence (DSM IV criteria) longer than 2 years
* asthma
* glaucoma
* pyloroduodenal obstruction (gastrointestinal stenosis)
* current pregnancy
* current breast feeding
* cardiac pacemaker
* heart or brain surgery
* metallic implants and alien objects in the body
* tattoos on head, neck or shoulders as well as permanent make-up
* claustrophobia

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-02-20 (Actual); Primary Completion 2019-05 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Number of participants with side effects | 1 year

SECONDARY OUTCOMES:
Performance differences in behavioral tasks after catecholamine depletion | 4 years
Differences in neural activation assessed during functional magnetic resonance imaging (fMRI) in the different conditions | 4 years
Differences in neural activation assessed during functional magnetic resonance imaging (fMRI) and in performance in behavioral tasks in the different conditions between the different genotypes | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Gregor Hasler, Prof. Dr. med, Principal Investigator — University Hospital of Psychiatry, University of Bern
Locations (1):
- University Hospital of Psychiatry, University of Bern, Bern, Switzerland

REFERENCES:
- [Background] Hasler G, Fromm S, Carlson PJ, Luckenbaugh DA, Waldeck T, Geraci M, Roiser JP, Neumeister A, Meyers N, Charney DS, Drevets WC. Neural response to catecholamine depletion in unmedicated subjects with major depressive disorder in remission and healthy subjects. Arch Gen Psychiatry. 2008 May;65(5):521-31. doi: 10.1001/archpsyc.65.5.521. PMID 18458204
- [Background] Grob S, Stern J, Gamper L, Moergeli H, Milos G, Schnyder U, Hasler G. Behavioral responses to catecholamine depletion in unmedicated, remitted subjects with bulimia nervosa and healthy subjects. Biol Psychiatry. 2015 Apr 1;77(7):661-7. doi: 10.1016/j.biopsych.2013.09.013. Epub 2013 Oct 25. PMID 24209774
- [Background] Homan P, Grob S, Milos G, Schnyder U, Hasler G. Reduction in total plasma ghrelin levels following catecholamine depletion: relation to bulimic and depressive symptoms. Psychoneuroendocrinology. 2013 Sep;38(9):1545-52. doi: 10.1016/j.psyneuen.2012.12.024. Epub 2013 Jan 16. PMID 23333252